CLINICAL TRIAL: NCT01973283
Title: Antidepressant Response in the Treatment of Depressive Symptoms and Frailty Characteristics in Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Patrick J. Brown, Associate Professor of Clinical Psychology (in Psychiatry), New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6470/7289R; K23MH099097-01A1 (NIH)
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Major Depressive Disorder; Dysthymic Disorder; Depressive Disorder, NOS
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Depression | interventions — Antidepressive Agents; Escitalopram; Duloxetine Hydrochloride; Open Abdomen Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medication Treatment (Experimental): Participants are treated with a flexible-dose antidepressant medication for a period of 8 weeks.
  Interventions: Drug: Antidepressant Medication

INTERVENTIONS:
Drug: Antidepressant Medication — If patient has a history of non-response or cannot tolerate escitalopram and/or duloxetine, then they will be treated openly with an approved antidepressant.
  Other Names: Escitalopram; Duloxetine; Open treatment

SUMMARY:
The goal of this open-administration treatment study of citalopram (or duloxetine) is to evaluate the effect of antidepressant medication on treating the syndrome of "frailty" in older adults with depressive symptoms. Patients with significant depressive symptoms (defined as CES-D (Center for Epidemiological Studies - Depression scale) > 10) and 1 or more symptoms of the frailty syndrome (exhaustion, decreased energy, weight loss, decreased grip strength, and slow/unsteady gait) will be evaluated and treated with citalopram (or duloxetine) for 8 weeks to test whether antidepressant medication improves both the syndrome of frailty and depressive symptoms. Patients evaluated at the Adult and Late Life Depression clinic and eligible to participate in the study will be treated with an antidepressant medication and assessed on the primary outcome variables (characteristics of frailty, depressive symptoms) as well as on secondary variables which include cognition (global cognition, episodic memory, executive function), and function (physical mobility, instrumental activities of daily living, and social functioning) prior to treatment initiation and following 8-weeks of treatment. The hypotheses for this protocol predict that we will discover a significant improvement on both frailty characteristics and depressive symptoms in this clinical population when treated with antidepressant medication (citalopram or duloxetine).

DETAILED DESCRIPTION:
Frailty, "a syndrome of decreased resiliency and reserves", is defined by five characteristics: 1)"shrinking" (definition: unintentional weight loss of > 10 lbs in prior year, or > 5% loss of body weight in prior year at follow-up), 2) weakness (definition: grip strength in lowest 20% at baseline, adjusted for gender and BMI), 3) poor endurance/energy (definition: self-report of exhaustion on 2 items on the CES-D), 4) slowness (definition: slowest 20% on timed 4 meter or 15 foot walk, adjusted for gender and standing height), and 5) low physical activity (definition: weighted score of kilocalories expended per week as calculated from the Minnesota Leisure Time Activity questionnaire). Frailty is associated with poor prognosis including hospitalization, falls, worsening disability and mobility, and death.

Data from the Cardiovascular Health Study document the rate of comorbid depressive symptoms in frail older adults (16.2% of older adults with at least 1 frailty characteristic had a CES-D > 10, including 31% of older adults with 3 or more frailty characteristics, compared to 2.6% of nonfrail older adults) despite study exclusion of individuals who were taking an antidepressant (this is in part why we chose to include patients with a CES-D of > 10, rather than requiring a diagnosis of a depressive disorder such as major depression or dysthymia for this study). The relationship between frailty and depression however goes beyond this association; the five defining characteristics of frailty (exhaustion, decreased energy, weight loss, decreased grip strength, and slow/unsteady gait) overlap significantly with symptoms of geriatric depression (decreased energy and motivation, psychomotor slowing, weight loss, decreased participation in leisure activities).

The proposed study is innovative in that it is focuses on a group of older adults who have been unrepresented (via exclusion criteria) in previous clinical studies (frail older adults with comorbid depressive symptoms), and it treats the comorbid depressive symptoms and targets characteristics of the frailty syndrome in the hopes of altering the prognostic trajectory of this clinical sample. This protocol serves two purposes: 1. It tests the feasibility of recruiting and retaining frail older adults with depressive symptoms in a treatment trial, and 2. It provides pilot data for the effectiveness of an antidepressant medication on treating the characteristics of frailty and the comorbid depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Anyone with 1 or more characteristics of frailty
* HRSD>16 and a DSM-IV depressive disorder (e.g. MDD, Dysthymia)
* Capable of providing informed consent
* Currently followed by a PCP (had an eval in last 6-months)

Exclusion Criteria:

* Acute cancer treatment
* Acute, severe or unstable medical illness
* End stage medical illness (e.g. liver, kidney, pulmonary)
* Mini Mental Exam < 24 or a diagnosis of dementia
* Individuals who do not have capacity to consent
* Diagnosis of substance abuse or dependence (last 12 months), excluding Nicotine dependence
* History of psychosis or psychotic disorder or bipolar disorder
* Patient is considered a significant risk of suicide
* Subject is considered based on history to be unlikely to respond to the single agent antidepressant (i.e., subjects with treatment resistant depression, including subjects with previous treatment with ECT)
* History of allergic or adverse reaction to escitalopram or duloxetine, or non-response to adequate trial of escitalopram (at least 4 weeks at dose of 20 mg) or duloxetine (at least 4 weeks at dose of 90mg).

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Brown, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Binder EF, Yarasheski KE, Steger-May K, Sinacore DR, Brown M, Schechtman KB, Holloszy JO. Effects of progressive resistance training on body composition in frail older adults: results of a randomized, controlled trial. J Gerontol A Biol Sci Med Sci. 2005 Nov;60(11):1425-31. doi: 10.1093/gerona/60.11.1425. PMID 16339329
- [Background] Brown M, Sinacore DR, Binder EF, Kohrt WM. Physical and performance measures for the identification of mild to moderate frailty. J Gerontol A Biol Sci Med Sci. 2000 Jun;55(6):M350-5. doi: 10.1093/gerona/55.6.m350. PMID 10843356
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Result] Brown PJ, Roose SP, O'Boyle KR, Ciarleglio A, Maas B, Igwe KC, Chung S, Gomez S, Naqvi M, Brickman AM, Rutherford BR. Frailty and Its Correlates in Adults With Late Life Depression. Am J Geriatr Psychiatry. 2020 Feb;28(2):145-154. doi: 10.1016/j.jagp.2019.10.005. Epub 2019 Oct 14. PMID 31734083
- [Result] Brown PJ, Ciarleglio A, Roose SP, Garcia CM, Chung S, Alvarez J, Stein A, Gomez S, Rutherford BR. Frailty Worsens Antidepressant Treatment Outcomes in Late Life Depression. Am J Geriatr Psychiatry. 2021 Sep;29(9):944-955. doi: 10.1016/j.jagp.2020.12.024. Epub 2020 Dec 25. PMID 33388223

RESULTS

PARTICIPANT FLOW:
Groups:
- Medication Treatment-8 Weeks: Participants are treated with a flexible-dose antidepressant medication for a period of 8 weeks.
  Antidepressant Medication: If patient has a history of non-response or cannot tolerate escitalopram and/or duloxetine, then they will be treated openly with an approved antidepressant.
Period: Overall Study
Arm/Group | Medication Treatment-8 Weeks
Started | 100
Completed | 96
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Medication Treatment
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.56 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 68
  More than one race | 5
  Unknown or Not Reported | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100
Hamilton Rating Scale for Depression (HRSD) [Mean (Standard Deviation); unit: Score on a scale] — Our target is depressive symptomatology as measured by the Hamilton Rating Scale for Depression (HRSD). The HRSD is a 24-item questionnaire used as an indication of depression and a guide to evaluating recovery. Total scores range from 0-74, not including atypical symptoms sub-scale. A score above 16 is typically considered to indicate the presence of depressive symptoms. Higher scores indicate greater severity.
  Score on a scale | 20.32 (5.84)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HRSD)
Description: Measure Description: Our target is depressive symptomatology as measured by the Hamilton Rating Scale for Depression (HRSD). The HRSD is a 24-item questionnaire used as an indication of depression and a guide to evaluating recovery. Total scores range from 0-74, not including atypical symptoms sub-scale. A score above 16 is typically considered to indicate the presence of depressive symptoms. Higher scores indicate greater severity.
Time Frame: Week 8
Population: Although 100 patients were assessed at baseline, 4 dropped out during the course of the 8-week trial. This leaves an analyzable sample of 96.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Treatment
Number analyzed (Participants) | 96
score on a scale | 13.3 (7.90)

2. Primary Outcome: Hamilton Rating Scale for Depression (HRSD)
Description: as for outcome 1
Time Frame: 6 Months
Population: Of the initial 100 patients assessed at baseline, 29 participants chose to not continue treatment past 8-weeks. As such, only 71 continued into the 10-month continuation phase of the project. Although these 29 were slightly older than the 71 who continued, they did not differ from those who continued in any other way including depression severity at baseline or 8-week treatment response. Because these 29 opted out of treatment after 8-weeks, only 71 were able to be analyzed at 6-months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Treatment
Number analyzed (Participants) | 71
score on a scale | 12.5 (7.44)

3. Primary Outcome: Hamilton Depression Rating Scale (HRSD)
Description: as for outcome 1
Time Frame: 12 Months
Population: Of the 71 who continued with treatment past 8-weeks, 11 dropped out between the 6- and 12-month assessment points. As such, 60 patients underwent 12-month assessments and were analyzable at 12-months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Treatment
Number analyzed (Participants) | 60
score on a scale | 13.6 (7.48)

4. Primary Outcome: Hamilton Depression Rating Scale: Stratified by Baseline Frailty
Description: as for outcome 1
Time Frame: Baseline (Week 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Frail: Participants who had 3 or more frailty characteristics (slow gait speed, weak grip strength, low physical activity levels, the presence of fatigue and significant weight loss, all determined using prespecified cut scores) at baseline are categorized as having frailty.
- Not/Intermediate Frail: Participants who had 0-2 frailty characteristics (slow gait speed, weak grip strength, low physical activity levels, the presence of fatigue and significant weight loss, all determined using prespecified cut scores) at baseline are categorized as either non-frail (0 characteristics) or intermediate frailty (1-2 characteristics).
Arm/Group | Frail | Not/Intermediate Frail
Number analyzed (Participants) | 49 | 51
score on a scale | 21 (6.61) | 19.7 (5.73)

5. Primary Outcome: Hamilton Depression Rating Scale: Stratified by Baseline Frailty
Description: as for outcome 1
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Frail | Not/Intermediate Frail
Number analyzed (Participants) | 48 | 48
score on a scale | 15.1 (8.23) | 11.6 (7.21)

6. Primary Outcome: Hamilton Depression Rating Scale: Stratified by Baseline Frailty
Description: as for outcome 1
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Frail | Not/Intermediate Frail
Number analyzed (Participants) | 31 | 40
score on a scale | 14.8 (8.65) | 10.8 (5.85)

7. Primary Outcome: Hamilton Depression Rating Scale: Stratified by Baseline Frailty
Description: as for outcome 1
Time Frame: Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Frail | Not/Intermediate Frail
Number analyzed (Participants) | 27 | 33
score on a scale | 14.3 (8.21) | 13.0 (6.91)

8. Secondary Outcome: World Health Organization Disability Assessment 2.0 (36-item)
Description: Assesses the level of functioning of patients, a component of the frailty evaluation. The scores assigned to each of the items: "none" (0), "mild" (1) "moderate" (2), "severe" (3), and "extreme" (4) - are summed. Each of the items is simply added up without recoding or collapsing of response categories; thus, there is no weighting of individual items. As a result, the simple sum of the scores of the items across all domains constitutes a statistic that is sufficient to describe the degree of functional limitations.
  Step 1 - Summing of recoded item scores within each domain. Step 2 - Summing of all six domain scores. Step 3 - Converting the summary score into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability).
Time Frame: Baseline (Week 0)
Population: Although 100 subjects enrolled in the study, only 12 subjects completed the baseline WHODAS assessment, so only 12 subjects' data were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Treatment
Number analyzed (Participants) | 12
score on a scale | 71.7 (24.8)

9. Secondary Outcome: World Health Organization Disability Assessment 2.0 (36-item)
Description: Assesses the level of functioning of patients, a component of the frailty evaluation. Simple: the scores assigned to each of the items - "none" (0), "mild" (1) "moderate" (2), "severe" (3), and "extreme" (4) - are summed. This method is referred to as simple scoring because the scores from each of the items are simply added up without recoding or collapsing of response categories; thus, there is no weighting of individual items. This approach is practical to use as a hand-scoring approach and may be the method of choice in busy clinical settings or in paper-pencil interview situations. As a result, the simple sum of the scores of the items across all domains constitutes a statistic that is sufficient to describe the degree of functional limitations.
  Step 1 - Summing of recoded item scores within each domain. Step 2 - Summing of all six domain scores. Step 3 - Converting the summary score into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability).
Time Frame: Week 8
Population: Although 100 subjects enrolled in the study, only 84 subjects completed the Week 8 WHODAS assessment, so only 84 subjects' data were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Treatment
Number analyzed (Participants) | 84
score on a scale | 68.7 (21.6)

10. Secondary Outcome: World Health Organization Disability Assessment 2.0 (36-item)
Description: as for outcome 8
Time Frame: 6 Months
Population: Although 100 subjects enrolled in the study, only 64 subjects completed the Month 6 WHODAS assessment, so only 64 subjects' data were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Treatment
Number analyzed (Participants) | 64
score on a scale | 66.7 (20.9)

11. Secondary Outcome: World Health Organization Disability Assessment 2.0 (36-item)
Description: as for outcome 8
Time Frame: 12 Months
Population: Although 100 subjects enrolled in the study, only 59 subjects completed the Month 12 WHODAS assessment, so only 59 subjects' data were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medication Treatment
Number analyzed (Participants) | 59
score on a scale | 67.8 (20.7)

12. Secondary Outcome: World Health Organization Disability Assessment 2.0 (36-item)--Stratified by Baseline Frailty
Description: as for outcome 8
Time Frame: Baseline (Week 0)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Frail | Not/Intermediate Frail
Number analyzed (Participants) | 7 | 5
score on a scale | 82.3 (24.1) | 56.8 (18.8)

13. Secondary Outcome: World Health Organization Disability Assessment 2.0 (36-item)--Stratified by Baseline Frailty
Description: as for outcome 8
Time Frame: Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Frail | Not/Intermediate Frail
Number analyzed (Participants) | 42 | 42
score on a scale | 77.9 (22.8) | 59.4 (15.8)

14. Secondary Outcome: World Health Organization Disability Assessment 2.0 (36-item)--Stratified by Baseline Frailty
Description: as for outcome 8
Time Frame: Month 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Frail | Not/Intermediate Frail
Number analyzed (Participants) | 29 | 35
score on a scale | 77.2 (19.9) | 58.0 (17.5)

15. Secondary Outcome: World Health Organization Disability Assessment 2.0 (36-item)--Stratified by Baseline Frailty
Description: as for outcome 8
Time Frame: Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Frail | Not/Intermediate Frail
Number analyzed (Participants) | 27 | 32
score on a scale | 80.9 (18.1) | 56.7 (15.8)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for 12 months
Arm/Group | Medication Treatment-8 Weeks
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 2/100
Other Adverse Events (participants affected / at risk) | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication Treatment-8 Weeks (N=100)
Fall (Injury, poisoning and procedural complications) | 2 (2) — Participants fell while standing or sitting and went to the emergency room for evaluation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT01973283/Prot_000.pdf
  • Informed Consent Form (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT01973283/ICF_001.pdf
  • Statistical Analysis Plan (2012-11-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT01973283/SAP_002.pdf